CLINICAL TRIAL: NCT00641394
Title: The Effect of Psychotherapy on Stress Biochemistry: A Randomized Blind Controlled Trial of Psychotherapy and Emotional Freedom Techniques (EFT)
Brief Title: The Effect of Psychotherapy on Stress Biochemistry: An RCT of Psychotherapy and Emotional Freedom Techniques (EFT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMI-CORT-32008
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Stress; Depression; Anxiety
Keywords: cortisol; hydrocortisone; psychotherapy; Emotional Freedom Techniques (EFT); Cognitive Behavioral Therapy (CBT); depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Psychotherapy: Emotional Freedom Techniques (EFT), a psychotherapy intervention with a somatic component
  Interventions: Behavioral: Psychotherapy: Emotional Freedom Techniques (EFT)
- 2 (Active Comparator): Psychotherapy: Cognitive Behavioral Therapy (CBT), a psychotherapy intervention
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- 3 (No Intervention)

INTERVENTIONS:
Behavioral: Psychotherapy: Emotional Freedom Techniques (EFT) — A form of therapy that includes cognitive reframing with somatic reinforcement through touch or tapping of specified points on the body
  Arms: 1
Behavioral: Cognitive Behavioral Therapy (CBT) — A form of therapy that focuses on negative cognitions of problems, and reframing them in positive terms, but without somatic reinforcement.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether there is a change in levels of cortisol, a key stress hormone, during the course of a psychotherapy session. The two forms of psychotherapy compared are Cognitive Behavioral Therapy (CBT) and Emotional Freedom Techniques (EFT). A no treatment control group provides a baseline measure. The change in cortisol level is compared between the start and end of a one hour session.

DETAILED DESCRIPTION:
Cortisol is a crucial physiological marker for stress. Stress produces elevated cortisol levels for as long as the body can supply the precursors. Elevated cortisol levels are associated with physical conditions such as impaired immune system function, cardiovascular disease, stroke, and accelerated aging. Elevated cortisol levels are also implicated in many psychological conditions. If the adrenal glands, which produce cortisol, are stimulated by the physical or psychological environment to produce stress hormones, they shunt production away from making DHEA, which is vital for cell regeneration.

The current pilot study examines the change in cortisol levels that result from a one hour psychotherapy session. It measures salivary cortisol, which indicates the levels of cortisol readily available to the body. This measure is relatively stable, and is not susceptible to large swings in the relatively brief period of a one hour psychotherapy session. Excluded are subjects with major depressive disorder, posttraumatic stress syndrome, and chronic diseases which have been shown to affect cortisol levels. Cortisol assessments will also take place in the afternoon or evening, to control for low waking cortisol which may be present in some normal subjects.

It is hypothesized that if psychotherapy is successful at treating trauma, cortisol levels will decline between the beginning of the hour and the end of the hour. The structure of the session is that the client discusses their emotional trauma in the first half of the session, and is treated with either cognitive behavioral therapy (CBT) or emotional freedom techniques (EFT) in the second half of the session. A no treatment control group provides baseline data. Half an hour is sufficient time for cortisol reuptake, and if therapy is successful at reducing physiological markers of stress, the client might demonstrate lower levels of cortisol at the conclusion of the psychotherapy session. Subjects who spontaneously have recall of a new significant trauma during the treatment portion of the session will also be excluded, since such recall can result in a cortisol spike. The study also evaluates a range of psychological conditions before and after the session using the SA-45. This brief questionnaire has subscales for anxiety, depression, phobias, hostility and other characteristics; these can be compared to cortisol levels to determine any correlations between psychological and physiological change.

ELIGIBILITY:
Inclusion Criteria:

* Good Health History

Exclusion Criteria:

* MDD (Major Depressive Disorder)
* PTSD (Post Traumatic Stress Disorder)
* Psychotropic Prescription Drug Use
* Currently Under Psychiatric Care
* Major disease, cancer, cardiovascular disease
* Autoimmune disease
* CFS (Chronic Fatigue Syndrome)
* Cushing's Syndrome
* Addison's Disease
* Spontaneous Trauma Recall in Final 20 minutes of Session
* History of Psychological Illness
* Pretest Cortisol level of .5 ng/ml or under, or 7 ng/ml or over

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
spot cortisol level | 60 minutes

SECONDARY OUTCOMES:
SA-45 symptom assessment questionnaire, with subscales for depression, anxiety, hostility, interpersonal sensitivity, phobias, and other psychological traits | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- [Result] Church D, Yount G, Brooks AJ. The effect of emotional freedom techniques on stress biochemistry: a randomized controlled trial. J Nerv Ment Dis. 2012 Oct;200(10):891-6. doi: 10.1097/NMD.0b013e31826b9fc1. PMID 22986277